CLINICAL TRIAL: NCT01904526
Title: Pharmacokinetic/Dynamic (PK/PD) Comparison of Guanfacine Extended Release (ER) and Immediate Release (IR) in Smokers
Brief Title: PK/PD Comparison of Guanfacine ER and IR
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Sherry McKee, Associate Professor of Psychiatry, Yale University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 1110009133; R01DA035001 (NIH); P50DA033945 (NIH)
Record Dates: First submitted 2013-07-12; First posted 2013-07-22 (Estimated); Results first posted 2018-04-23 (Actual); Last update posted 2020-03-06 (Actual); Status verified 2020-03

CONDITIONS: Smoking
Keywords: Guanfacine; PK/PD; Smokers
MeSH Terms: conditions — Smoking | interventions — Guanfacine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Guanfacine (Experimental): Guanfacine 3 mg/day immediate release followed by Guanfacine 4mg/day extended release followed by Guanfacine 6 mg/day extended release
  Interventions: Drug: Guanfacine

INTERVENTIONS:
Drug: Guanfacine — 3mg/day IR with 3-week lead-in period. Maintained at steady state to complete lab session. After completion of lab session, 1-week lead-in medication period to 4mg/day ER. Maintained at steady state to complete lab session. After completion of lab session, 1-week lead-in medication period to 6mg/day ER. Maintained at steady state to complete lab session. 5-day taper after lab.
  Other Names: Tenex; Intuniv

SUMMARY:
Evaluate whether a 4mg/day or 6/mg day dose of extended-release guanfacine produces pharmacokinetic/dynamic (PK/PD) properties similar to 3mg/day immediate release guanfacine.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65
* Able to read, write and comprehend English
* Smoker
* Able to take oral medications and willing to adhere to medication regimen
* Provide evidence of a stable living residence in the last 2 months, have reasonable transportation to the study site, and have no plans to move within the next 3 months or unresolved legal problems.

Exclusion Criteria:

* Any significant current medical conditions that would contraindicate smoking
* Current Diagnostic and Statistical Manual of Mental Disorders (DSM-IV) abuse or dependence of other substances, other than nicotine dependence or alcohol abuse
* Positive test results at intake appointment on urine drug screens for illicit drugs
* Past 30 day use of psychoactive drugs including anxiolytics and antidepressants
* Women who are pregnant or nursing
* Suicidal, homicidal or evidence of current mental illness such as schizophrenia, bipolar disorder or major depression, or anxiety disorders
* Meeting DSM-IV criteria for current attention deficit hyperactivity disorder (ADHD)
* Individuals who are currently taking medications known to be effective for smoking cessation or are regular users of other tobacco products in the past 30 days
* Only one member per household can participate in the study
* Specific exclusions for administration of guanfacine not already specified include:

  * EKG evidence at baseline screening of any clinically significant conduction abnormalities or arrhythmias
  * Known intolerance for guanfacine or any alpha blocker
  * History of fainting, syncopal attacks
  * Heart failure or myocardial infarction
  * Impaired liver (as indicated by aspartate aminotransferase (AST), alanine aminotransferase (ALT) >3x normal)
  * Renal function (as indicated by estimated creatinine clearance <60cc/min)
  * Treatment with any antihypertensive drug or any alpha-adrenergic blocker
  * Use of any central nervous system depressant (e.g., phenothiazines, barbiturates, benzodiazepines)
  * Use of strong cytochrome P450 3A4 (CYP3A4) inhibitors (e.g., ketoconazole) or inducers (e.g., rifampin), or consumption of grapefruit juice
* Subjects may have not donated blood in the past 8 weeks or have been involved in other investigational studies that involve substantial blood draws or medications unknown to us

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2013-07; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sherry A McKee, PhD, Principal Investigator — Yale University
Locations (1):
- Yale Center for Clinical Investigations, Yale University, New Haven, Connecticut, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Guanfacine: Guanfacine: 3mg/day immediate release (IR) with 3-week lead-in period. Maintained at steady state to complete lab session. After completion of lab session, 1-week lead-in medication period to 4mg/day extended release (ER). Maintained at steady state to complete lab session. After completion of lab session, 1-week lead-in medication period to 6mg/day ER. Maintained at steady state to complete lab session. 5-day taper after lab.
Period: Overall Study
Arm/Group | Guanfacine
Started | 5
Completed | 5
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Guanfacine
Number analyzed (Participants) | 5
Age, Continuous [Mean (Standard Deviation); unit: Years] | 45.8 (2.49)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 3

OUTCOME MEASURES:

1. Primary Outcome: Plasma Trough Levels of Guanfacine
Description: Evaluate whether a 4mg/day or 6mg/day dose of extended-release guanfacine produces pharmacokinetic (PK) properties similar to 3mg/day immediate release guanfacine by measuring plasma trough levels of guanfacine for each dose
Time Frame: +24 hours on Lab Session days (Days 22, 49, 58)
Population: 3 mg/day IR (Day 22) followed by 4mg/day ER (Day 49) followed by 6mg/day ER (Day 58)
Measure: Mean (Standard Error); unit: ng/ml
Groups:
- Guanfacine 3mg/Day Immediate Release: Guanfacine: 3mg/day immediate release
- Guanfacine 4mg/Day Extended Release: Guanfacine: 4mg/day extended release
- Guanfacine 6mg/Day Extended Release: Guanfacine: 6mg/day extended release
Arm/Group | Guanfacine 3mg/Day Immediate Release | Guanfacine 4mg/Day Extended Release | Guanfacine 6mg/Day Extended Release
Number analyzed (Participants) | 5 | 5 | 5
ng/ml | 3.40 (0.33) | 3.46 (0.67) | 5.92 (1.02)

2. Secondary Outcome: Heart Rate
Description: Evaluate the safety and tolerability of guanfacine by measuring physiologic reactivity (e.g., heart rate)
Time Frame: Last day of titration period 1 (Day 21) to the last day of titration period 3 (Day 57)
Population: Last day of titration period: 3 mg/day IR (Day 21) followed by 4mg/day ER (Day 48) followed by 6mg/day ER (Day 57)
Measure: Mean (Standard Error); unit: beats per minute
Arm/Group | Guanfacine 3mg/Day Immediate Release | Guanfacine 4mg/Day Extended Release | Guanfacine 6mg/Day Extended Release
Number analyzed (Participants) | 5 | 5 | 5
beats per minute | 59.6 (1.75) | 58.8 (3.97) | 61.6 (5.30)

3. Secondary Outcome: Systolic Blood Pressure
Description: Evaluate the safety and tolerability of guanfacine by measuring physiologic reactivity (e.g., systolic blood pressure)
Time Frame: Last day of titration period 1 (Day 21) to the last day of titration period 3 (Day 57)
Population: Last day of titration period: 3 mg/day IR (Day 21) followed by 4 mg/kg ER (Day 48) followed by 6 mg/day ER (Day 57)
Measure: Mean (Standard Error); unit: mmHg
Arm/Group | Guanfacine 3mg/Day Immediate Release | Guanfacine 4mg/Day Extended Release | Guanfacine 6mg/Day Extended Release
Number analyzed (Participants) | 5 | 5 | 5
mmHg | 101.0 (3.73) | 107.4 (7.51) | 108.4 (7.16)

ADVERSE EVENTS:
Arm/Group | Guanfacine 3mg/Day Immediate Release | Guanfacine 4mg/Day Extended Release | Guanfacine 6mg/Day Extended Release
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/5 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/5 | 0/5
Other Adverse Events (participants affected / at risk) | 3/5 | 4/5 | 4/5
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Guanfacine 3mg/Day Immediate Release (N=5) | Guanfacine 4mg/Day Extended Release (N=5) | Guanfacine 6mg/Day Extended Release (N=5)
Dry mouth (General disorders) | 2 | 4 | 4
Drowsiness (General disorders) | 3 | 3 | 3
Dizziness (General disorders) | 2 | 2 | 2
Constipation (Gastrointestinal disorders) | 2 | 2 | 2
Fatigue (General disorders) | 3 | 3 | 3
Headache (General disorders) | 2 | 1 | 0
Insomnia (General disorders) | 0 | 1 | 0
Gas pains (Gastrointestinal disorders) | 2 | 2 | 3
Diarrhea (Gastrointestinal disorders) | 1 | 0 | 0
Loss of appetite (General disorders) | 1 | 0 | 1
Runny nose (General disorders) | 1 | 0 | 1
Weakness (General disorders) | 1 | 0 | 2
Nausea/vomiting (General disorders) | 0 | 0 | 0
Chest pain (Cardiac disorders) | 1 | 0 | 0
Shortness of breath (General disorders) | 0 | 0 | 0
Skin rash (General disorders) | 0 | 0 | 0
Swelling of hands or feet (General disorders) | 0 | 0 | 0
Blurred vision (General disorders) | 0 | 0 | 0
Yellowing of the eyes or skin (General disorders) | 0 | 0 | 0
Mental/mood changes (General disorders) | 0 | 0 | 0
Tingling of the hands or feet (General disorders) | 0 | 0 | 0
Impotence (General disorders) | 2 | 0 | 1
Decreased sexual desire (General disorders) | 1 | 0 | 1
Vision changes (General disorders) | 0 | 0 | 0
Taste changes (General disorders) | 1 | 1 | 1
Ringing in ears (General disorders) | 1 | 1 | 1
Leg cramps (General disorders) | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No